CLINICAL TRIAL: NCT01368913
Title: MINRIN® Orally Disintegrating Tablet (Fast Dissolving Desmopressin) and Tablets in Treatment of Primary Nocturnal Enuresis With Special Focus on Patient Satisfaction
Brief Title: MINRIN® Orally Disintegrating Tablet (Fast Dissolving Desmopressin) and Tablets in Treatment of Primary Nocturnal Enuresis
Acronym: MELT
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Collaborators: Ferring Arzneimittel GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 000018
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients treated with orally disintegrating tablet
- Patients treated with tablets

SUMMARY:
Desmopressin in treatment of nocturnal enuresis (bedwetting).

ELIGIBILITY:
Inclusion Criteria:

* Treatment of primary nocturnal enuresis within an overall therapeutical concept, eg, in cases of failure of other non-medicinal therapies or with indication of a medicinal therapy caused by nocturnal ADH deficiency
* The patients and their parents have been informed about the study and have given their written consent for participation.

Exclusion Criteria:

* The prescription of Minirin® tablets / Minirin® orally disintegrating tablet (fast dissolving desmopressin) is contraindicated

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary nocturnal enuresis
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2011-06; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assessment of patient and parent satisfaction | 3 months

SECONDARY OUTCOMES:
Number of wet nights | 3 months
Assessment of drinking volume | 3 months
Assessment of urine volume | 3 months
Assessment of patient compliance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (73):
- Germany (73):
  - Investigational Site, Bad Bergzaben
  - Investigational Site, Kaiserdamm 26, Berlin
  - Investigational Site, Mahlsdorfer Straße 39-40, Berlin
  - Investigational Site, Neckarstrasse 7, Berlin
  - Investigational Site, Potsdamer Chussee 80, Berlin
  - Investigational Site, Bingen
  - Investigational Site, Zossener Damm 42, Blankenfelde
  - Investigational Site , An der Ziegelei 8, Bonn
  - Investigational Site, Reichsstraße 51, Bonn
  - Investigational Site, Brackenheim
  - Investigational Site, Brunsbüttel
  - Investigational Site, Cologne
  - Investigational Site, Crailsheim
  - Investigational Site, Dresden
  - Investigational Site, Duisburg
  - Investigational Site, Suitberutsstraße 31, Düsseldorf
  - Investigational Site, Westfalenstraße 26, Düsseldorf
  - Investigational Site, Düsseldorf
  - Investigational Site, Erfurt
  - Investigational Site, Espelkamp
  - Investigational Site, Ettenheim
  - Investigational Site, Forchheim
  - Investigational Site, Frankfurt am Main
  - Investigational Site, Friedberg
  - Investigational Site, Fulda
  - Investigational Site, Gelsenkirchen
  - Investigational Site, Germering
  - Investigational Site, Gernsbach
  - Investigational Site, Gilching
  - Investigational Site, Görlitz
  - Investigational Site, Groß-Umstadt
  - Investigational Site, Großenhain
  - Investigational Site, Großröhrsdorf
  - Investigational Site, Hammelburg
  - Investigational Site, Hanover
  - Investigational Site, Harsewinkel-Greffen
  - Investigational Site, Homburg/Saar
  - Investigational Site, Hürth
  - Investigational Site, Hüttenberg
  - Investigational Site, Itzehoe
  - Investigational Site, Karlsruhe
  - Medical Faculty of University Clinic - Schwanenweg 20, Kiel
  - Investigational Site, Königswinter-Oberpl.
  - Investigational Site, Neue Linner Straße 77, Krefeld
  - Investigational Site, Langerwehe
  - Investigational Site, Lehrte
  - Investigational Site, Lengerich
  - Investigational Site, Leverkusen-Schlebusch
  - Investigational Site, Minden
  - Investigational Site, Mönchengladbach
  - Investigational Site, Mutzschen
  - Investigational Site, Neu Wulmstorf
  - Investigational Site, Neumünster
  - Investigational Site, Oberhausen
  - Investigational Site, Oederan
  - Investigational Site, Waldstraße 43, Offenbach
  - Investigational Site, Offenbach
  - Investigational Site, Oldenburg
  - Investigational Site, Ottobrunn bei München
  - Investigational Site, Potsdam
  - Investigational Site, Rothenburg
  - Investigational Site, Rottweil
  - Investigational Site, Rüsselsheim am Main
  - Investigational Site, Schopfheim
  - Investigational Site, Schwabach
  - Investigational Site, Strausberg
  - Investigational Site, Traunstein
  - Investigational Site, Trittau
  - Investigational Site, Varel
  - Investigational Site, Wertheim am Main
  - Investigational Site, Wiefelstede
  - Investigational Site, Wilkau-Haßlau
  - Investigational Site, Wuppertal